CLINICAL TRIAL: NCT07012395
Title: Phase 2 Platform Trial to Assess the Efficacy and Safety of Long-acting Antibodies as Single Agents and in Combinations for Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study of Long-acting Antibodies Alone and in Combinations for Moderate to Severe Ulcerative Colitis
Acronym: SKYLINE-UC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Spyre Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPY123-201
Record Dates: First submitted 2025-05-27; First posted 2025-06-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Diseases; Colitis; Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases; Colitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Intervention Specific Appendix - SPY001: Part A (Experimental): Participants will receive open-label dose of SPY001
  Interventions: Drug: SPY001
- Intervention Specific Appendix - SPY002: Part A (Experimental): Participants will receive open-label dose of SPY002
  Interventions: Drug: SPY002
- Intervention Specific Appendix - SPY003: Part A (Experimental): Participants will receive open-label dose of SPY003
  Interventions: Drug: SPY003
- Intervention Specific Appendix - SPY001 Dosing Regimen 1: Part B (Experimental): Participants will receive double-blind dosing regimen 1 of SPY001
  Interventions: Drug: SPY001
- Intervention Specific Appendix - SPY001 Dosing Regimen 2: Part B (Experimental): Participants will receive double-blind dosing regimen 2 of SPY001
  Interventions: Drug: SPY001
- Intervention Specific Appendix - SPY002 Dosing Regimen 1: Part B (Experimental): Participants will receive double-blind dosing regimen 1 of SPY002
  Interventions: Drug: SPY002
- Intervention Specific Appendix - SPY002 Dosing Regimen 2: Part B (Experimental): Participants will receive double-blind dosing regimen 2 of SPY002
  Interventions: Drug: SPY002
- Intervention Specific Appendix - SPY003 Dosing Regimen 1: Part B (Experimental): Participants will receive double-blind dosing regimen 1 of SPY003
  Interventions: Drug: SPY003
- Intervention Specific Appendix - SPY003 Dosing Regimen 2: Part B (Experimental): Participants will receive double-blind dosing regimen 2 of SPY003
  Interventions: Drug: SPY003
- Intervention Specific Appendix - SPY120: Part B (Experimental): Participants will receive double-blind dose of SPY001 and SPY002
  Interventions: Drug: SPY001; Drug: SPY002
- Intervention Specific Appendix - SPY130: Part B (Experimental): Participants will receive double-blind dose of SPY001 and SPY003
  Interventions: Drug: SPY001; Drug: SPY003
- Intervention Specific Appendix - SPY230: Part B (Experimental): Participants will receive double-blind dose of SPY002 and SPY003
  Interventions: Drug: SPY002; Drug: SPY003
- Placebo: Part B (Placebo Comparator): Participants will receive matching placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SPY001 — Experimental
  Other Names: SPY001-001
  Arms: Intervention Specific Appendix - SPY001 Dosing Regimen 1: Part B; Intervention Specific Appendix - SPY001 Dosing Regimen 2: Part B; Intervention Specific Appendix - SPY001: Part A; Intervention Specific Appendix - SPY120: Part B; Intervention Specific Appendix - SPY130: Part B
Drug: SPY002 — Experimental
  Other Names: SPY002-091
  Arms: Intervention Specific Appendix - SPY002 Dosing Regimen 1: Part B; Intervention Specific Appendix - SPY002 Dosing Regimen 2: Part B; Intervention Specific Appendix - SPY002: Part A; Intervention Specific Appendix - SPY120: Part B; Intervention Specific Appendix - SPY230: Part B
Drug: SPY003 — Experimental
  Other Names: SPY003-207
  Arms: Intervention Specific Appendix - SPY003 Dosing Regimen 1: Part B; Intervention Specific Appendix - SPY003 Dosing Regimen 2: Part B; Intervention Specific Appendix - SPY003: Part A; Intervention Specific Appendix - SPY130: Part B; Intervention Specific Appendix - SPY230: Part B
Other: Placebo — Placebo
  Arms: Placebo: Part B

SUMMARY:
This is a Phase 2, multicenter, proof-of-concept platform study in adult participants with moderately to severely active ulcerative colitis (UC). The primary goal of the study is to assess the efficacy and safety of multiple interventions following intravenous (IV) induction and subcutaneous (SC) maintenance treatment.

DETAILED DESCRIPTION:
This platform study will evaluate the efficacy and safety of investigational treatments, including 3 monotherapies and 3 combination therapies, for moderately to severely active UC in adults. The study will progress in two parts.

Part A is the open-label portion of the study assessing safety and preliminary efficacy of monotherapies.

Part B, which will be open for enrollment after Part A, is the randomized, placebo-controlled portion of the study assessing the safety and efficacy of the 6 interventions (3 monotherapies and 3 combinations) compared to placebo.

Intervention arms will be added to the study over time and may complete at different times.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of UC for ≥3 months before Day 1, confirmed by endoscopy and histology either previously or during Screening
* Active UC with disease extent of ≥15 cm from the anal verge, as confirmed by Screening endoscopy (up to approximately 15% allowed to have only proctitis)
* Moderately to severely active disease as defined by a modified Mayo score of 5-9, rectal bleeding subscore of ≥1, and Mayo endoscopic subscore ≥2

Exclusion Criteria:

* Current diagnosis of Crohn's disease or Inflammatory Bowel Disease (IBD)-Undefined
* Confirmed or suspected fulminant colitis, toxic megacolon, bowel perforation and/or other conditions that will likely require surgery during induction
* Failed 4 or more approved or investigational advanced therapy classes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 645 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Part A: Change in Robarts Histopathology Index (RHI) | Week 12
  Change in Robarts Histopathology Index (RHI) from baseline at Week 12 will be assessed. The RHI is used to quantify and assess histological activity of UC, comprising of scores for inflammatory infiltrates, neutrophils, erosions or ulceration. Scores are assigned to each of these features, with a total ranging from 0 (no disease activity) to 33 (most severe disease activity). Higher score indicates more severe disease.
Part B: Percentage of participants with clinical remission | Week 12
  Percentage of participants with clinical remission at Week 12 will be assessed. Clinical remission is based on the modified Mayo subscores, which consist of a rectal bleeding subscore (ranging from 0 to 3), stool frequency subscore (ranging from 0 to 3), and endoscopic subscore (ranging from 0 to 3), as assessed by central reading. Higher scores indicate more severe disease.

SECONDARY OUTCOMES:
Part A: Percentage of participants with clinical remission | Week 12
  Percentage of participants with clinical remission at Week 12 will be assessed. Clinical remission is based on the modified Mayo subscores, which consist of a rectal bleeding subscore (ranging from 0 to 3), stool frequency subscore (ranging from 0 to 3), and endoscopic subscore (ranging from 0 to 3), as assessed by central reading. Higher scores indicate more severe disease.
Part A: Percentage of participants with endoscopic improvement | Week 12
  Percentage of participants with endoscopic improvement at Week 12 will be assessed. Endoscopic improvement based on the Mayo endoscopic subscore (ranging from 0 to 3), as assessed by central reading. Higher score indicates more severe disease.
Part B: Percentage of participants with endoscopic improvement | Week 12
  Percentage of participants with endoscopic improvement at Week 12 will be assessed. Endoscopic improvement based on the Mayo endoscopic subscore (ranging from 0 to 3), as assessed by central reading. Higher score indicates more severe disease.
Part B: Percentage of participants with clinical response | Week 12
  Percentage of participants with clinical response at Week 12 will be assessed. Clinical response is based on the modified Mayo Score, which consist of a rectal bleeding subscore (ranging from 0 to 3), stool frequency subscore (ranging from 0 to 3), and endoscopic subscore (ranging from 0 to 3), as assessed by central reading. Higher scores indicate more severe disease.
Part B: Percentage of participants with histologic improvement | Week 12
  Percentage of participants with histologic improvement at Week 12 will be assessed. Histologic improvement is based on the Geboes score. The Geboes histologic index includes 7 histological features (architectural change, chronic inflammatory infiltrate, lamina propria neutrophils and eosinophils, neutrophils in epithelium, crypt destruction and erosion or ulcers). The Geboes score has 6 grades from 0 to 5, with each grade of the score divided into 4 or 5 subcategories; the score ranges from 0.0 to 5.4. Higher score indicates more severe disease.
Part B: Percentage of participants achieving histologic endoscopic mucosal improvement (HEMI). | Week 12
  Percentage of participants with HEMI at Week 12 will be assessed. Mucosal improvement is based on the Mayo endoscopic subscore and the Geboes score. The Mayo endoscopic subscore ranges from 0 to 3, as assessed by central reading. Higher score indicates more severe disease. The Geboes histologic index includes 7 histological features (architectural change, chronic inflammatory infiltrate, lamina propria neutrophils and eosinophils, neutrophils in epithelium, crypt destruction and erosion or ulcers). The Geboes score has 6 grades from 0 to 5, with each grade of the score divided into 4 or 5 subcategories; the score ranges from 0.0 to 5.4. Higher score indicates more severe disease
Part B: Percentage of participants with clinical remission | Week 48
  Percentage of participants with clinical remission at Week 48 will be assessed. Clinical remission is based on the modified Mayo subscores, which consist of a rectal bleeding subscore (ranging from 0 to 3), stool frequency subscore (ranging from 0 to 3), and endoscopic subscore (ranging from 0 to 3), as assessed by central reading. Higher scores indicate more severe disease.

CONTACTS AND LOCATIONS:
Overall Officials: SKYLINE-UC Study Director, Study Director — Spyre Therapeutics
Locations (101):
- United States (19):
  - Site 024, Canoga Park, California
  - Site 012, Lancaster, California
  - Site 033, Colorado Springs, Colorado
  - Site 007, Kissimmee, Florida
  - 029, Miami, Florida
  - Site 006, Kansas City, Kansas
  - Site 035, Marrero, Louisiana
  - Site 011, Glen Burnie, Maryland
  - Site 003, Boston, Massachusetts
  - 040, Chapel Hill, North Carolina
  - Site 016, Winston-Salem, North Carolina
  - Site 025, Providence, Rhode Island
  - Site 017, Kingsport, Tennessee
  - Site 013, Cedar Park, Texas
  - Site 005, Garland, Texas
  - Site 002, San Antonio, Texas
  - Site 008, Southlake, Texas
  - Site 009, Webster, Texas
  - Site 019, Tacoma, Washington
- Australia (3):
  - Site 202, Heidelberg
  - Site 204, Liverpool
  - Site 207, Woolloongabba
- Bosnia and Herzegovina (3):
  - Site 481, Banja Luka
  - Site 484, Mostar
  - Site 483, Sarajevo
- Canada (3):
  - Site 083, London, Ontario
  - Site 085, Greater Sudbury
  - Site 086, London
- Site 531, Brno, Czechia
- Georgia (10):
  - Site 584, Kutaisi
  - Site 589, Marneuli
  - Site 581, Tbilisi
  - Site 588, Tbilisi
  - Site 583, Tbilisi
  - Site 586, Tbilisi
  - Site 582, Tbilisi
  - Site 587, Tbilisi
  - Site 590, Tbilisi
  - Site 585, Tbilisi
- Site 604, Berlin, Germany
- Israel (5):
  - Site 445, Beer Yaaqov
  - Site 441, Beersheba
  - Site 443, Haifa
  - Site 444, Jerusalem
  - Site 446, Jerusalem
- Moldova (5):
  - Site 713, Chisinau
  - Site 711, Chisinau
  - Site 712, Chisinau
  - Site 714, Chisinau
  - Site 715, Chisinau
- Poland (9):
  - Site 735, Katowice
  - Site 737, Szczecin
  - Site 733, Szczecin
  - Site 739, Warsaw
  - Site 731, Warsaw
  - Site 750, Warsaw
  - Site 738, Wroclaw
  - Site 734, Wroclaw
  - Site 747, Wroclaw
- Serbia (7):
  - Trial Site 804, Belgrade
  - Site 802, Belgrade
  - Site 807, Belgrade
  - Site 803, Belgrade
  - Site 805, Niš
  - Site 806, Užice
  - Site 801, Zrenjanin
- South Korea (12):
  - Site 357, Busan
  - Site 354, Daegu
  - Site 358, Daegu
  - Site 361, Daegu
  - Site 355, Daejeon
  - Site 356, Seoul
  - Site 351, Seoul
  - Site 352, Seoul
  - Site 360, Seoul
  - Site 362, Seoul
  - Site 359, Suwon
  - Site 353, Wŏnju
- Spain (3):
  - Site 834, Madrid
  - Site 837, Madrid
  - Site 836, Ourense
- Switzerland (3):
  - Site 852, Basel
  - Site 853, Bern
  - Site 851, Sankt Gallen
- Taiwan (4):
  - Site 394, Changhua
  - Site 392, Chiayi City
  - Site 396, Taichung
  - Site 391, Taipei
- Ukraine (13):
  - Site 906, Ivano-Frankivsk
  - Site 902, Kyiv
  - Site 904, Kyiv
  - Site 905, Kyiv
  - Site 913, Kyiv
  - Site 911, Kyiv
  - Site 903, Kyiv
  - Site 901, Lutsk
  - Site 909, Lviv
  - Site 912, Lviv
  - Site 914, Poltava
  - Site 908, Vinnytsia
  - Site 907, Vinnytsia

IPD SHARING:
Plan to Share IPD: No